CLINICAL TRIAL: NCT03645824
Title: A Phase II Trial in Patients With Myelofibrosis (Primary, Post-ET or Post PV-MF) Treated With the Selective JAK2 Inhibitor Pacritinib Before Reduced-intensity Conditioning Allogeneic Stem Cell Transplantation
Brief Title: Myelofibrosis Treated With Pacritinib Before aSCT. (HOVON134MF)
Acronym: HOVON134MF
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: Dutch Cancer Society (Other); CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO134; 2015-000195-98 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-08-24 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Myelofibrosis
Keywords: Hemato-Oncology; Allogeneic Stem Cell Transplantation; Pacritinib; JAK2 inhibitor; Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pacritinib treatment befor allo-SCT (Experimental): The effect of pacritinib treatment during 3 to 4 cycles before allo-SCT on engraftment 6 months (day +180) post allo-SCT in MF patients.
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Patients receive up to 4 cycles of pacritinib before allo-SCT

SUMMARY:
The only curative treatment for patients with myelofibrosis (MF) is allogeneic stem cell transplantation (SCT). Treatment with JAK2 inhibitors like pacritinib improves condition of MF patients, decreases spleen size and might diminish graft-versus-host disease (GvHD), thereby improving the outcome of SCT.

DETAILED DESCRIPTION:
Despite recent new therapeutic options, allogeneic Stem Cell Transplantation remains the only curative option in patients with Myelofibrosis. Therefore, optimalization of this therapy remains a major challenge. Improvement of the clinical condition of these patients, decreasing spleen size can be accomplished by JAK2 inhibitor treatment and might improve SCT outcome. In addition, selective JAK2 inhibitors might modulate GvHD which can also add to improved SCT outcome. Also, decreasing the burden/activity of the disease before allo-SCT might also improve final disease response. The first, limited, clinical data of ruxolitinib treatment before allo-SCT show controversial effects on the outcome of SCT. Therefore, additional prospective clinical trials have to be done to establish the role of JAK2 inhibition before allogeneic SCT. Since ruxolitinib has considerable myelosuppressive effects which might limit the clinical use in some MF patients, other selective JAK2 inhibitors might be useful in this setting. Pacritinib, as a JAK2/FLT3 inhibitor, has a very potent JAK2 inhibitory activity without myelosuppressive effects and might therefore be more suitable than ruxolitinib. The major possible side effects are gastro-intestinal and can be managed with medication. In several studies, pacritinib has shown to be effective in decreasing spleen size and has shown to improve clinical condition of patients. Therefore, this compound seems promising in improving the outcome of allo-SCT. Although pacritinib causes no inhibition of JAK1 activity and therefore might have limited effects in decreasing inflammatory response, this might also be of benefit since a "withdrawal syndrome" as has been described after cessation of ruxolitinib is not to be expected.

With this trial, using pacritinib treatment before allo-SCT, the issue of improvement of SCT outcome will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of post-ET, post-PV or primary myelofibrosis
* Intermediate-2 or high-risk according to DIPSS plus (Appendix E)
* Age 18-70 years inclusive
* WHO performance status 0-2 (Appendix C)
* All men and women of childbearing potential must agree to use adequate contraception during the study
* Written informed consent
* Patient is capable of giving informed consent

Exclusion Criteria:

* Previous treatment with JAK2 inhibitors within 2 weeks of study inclusion. Patients who have been treated with pacritinib as their previous JAK2 inhibitor treatment cannot participate in this study
* Any GI or metabolic condition (e.g. inflammatory or chronic functional bowel disorder such as Crohn's Disease, Inflammatory Bowel Disease, chronic diarrhea or constipation) that could interfere with absorption of oral medication
* Left ventricular cardiac ejection fraction of ≤ 45% by echocardiogram or multigated acquisition (MUGA) scan
* Impaired liver and renal function, defined by liver transaminases (aspartate aminotransferase [AST]/serum glutamic oxaloacetic transaminase [SGOT] and alanine aminotransferase [ALT]/serum glutamic pyruvic transaminase [SGPT]), >3 × the upper limit of normal (ULN) (AST/ALT >5 × ULN if transaminase elevation is related to MF), direct bilirubin >4× ULN, and creatinine clearance ˂ 40 ml/min.
* Impaired coagulation function, defined by prothrombin time (PT)/international normalized ratio (INR), partial thromboplastin time (APTT)>1.5 x ULN.
* Experimental treatment within four weeks before inclusion for PMF, Post-PV, or Post-ET MF
* Severe pulmonary dysfunction (CTCAE grade III-IV, see appendix D)
* Treatment with a potent strong CYP3A4 inhibitor or a strong cytochrome P450 (CYP450) inducer within the last 2 weeks
* Treatment with anticoagulation or antiplatelet agents, except for aspirin dosages of ≤100 mg per day, within the last 2 weeks
* New York Heart Association Class II, III, or IV congestive heart failure
* QTc prolongation >450 ms as assessed by ECG and corrected by Federicia method or other factors that increase the risk for QT interval prolongation (e.g., heart failure, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], family history of long QT interval syndrome, or concomitant use of medications that may prolong QT interval)
* Significant recent bleeding history defined as NCI CTCAE grade ≥2 within the last 3 months, unless precipitated by an inciting event (e.g., surgery, trauma, injury)
* Any history of CTCAE grade ≥2 non-dysrhythmia cardiac conditions within the last 6 months. Patients with asymptomatic grade 2 non-dysrhythmia cardiac conditions may be considered for inclusion, with the approval of the principal investigator, if stable and unlikely to affect patient safety.
* Any history of CTCAE grade ≥2 cardiac dysrhythmias within the last 6 months. Patients with non-QTc CTCAE grade 2 cardiac dysrhythmias may be considered for inclusion, with the approval of the principal investigator, if the dysrhythmias are stable, asymptomatic, and unlikely to affect patient safety.
* Patients with active, uncontrolled infections
* Patients known to be HIV (human immunodeficiency virus)-positive
* Active hepatitis A, B or C
* History of active malignancy during the past 3 years, except basal carcinoma of the skin or stage 0 cervical carcinoma
* Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, cancer, etc.)
* Pregnant or breastfeeding women
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving allo-SCT, with failure within or at day 180 post-transplant. | 2 years
  Failure can be defined by one of the following parameters:
  * Primary graft failure
  * Acute graft versus host disease grade 3-4
  * Secondary graft failure
  * Death, from any cause

SECONDARY OUTCOMES:
Adverse events | 5 years
  Adverse events will be monitored.
Progression free survival | 5 years
  Progression free survival as time between registration or SCT until progression/relapse or death from any cause
Overall survival | 5 years
  Over all survival, calculated from either registration or SCT.
Relapse mortality | 5 years
  Death due to the disease or after progression
Non-relapse mortality | 5 years
  Death not due to disease or relapse
Quality of life during and after treatment | 5 years
  Quality of life during and after treatment will be recorded by use of the MPN-SAF questionnaire.
  From a total of 27 questions, the scores (from 0 to 10) from the following 10 questions are added and subsequently averaged to come to a total quality of life score.
  * fatigue
  * satisfction after a meal
  * stomach complaints
  * not able to perform activities
  * concentration problems
  * night sweat
  * itch
  * bone pain
  * fever
  * sudden weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Peter AW te Boekhorst, M.D. PhD, Principal Investigator — Erasmus Medical Center
Locations (12):
- Belgium (4):
  - BE-Antwerpen-ZNASTUIVENBERG, Antwerp
  - BE-Gent-UZGENT, Ghent
  - BE-Leuven-UZLEUVEN, Leuven
  - BE-Roeselare-AZDELTA, Roeselare
- Netherlands (8):
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Groningen-UMCG, Groningen
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-EMCDANIEL, Rotterdam
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Utrecht-UMCUTRECHT, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HOVON Foundation (STICHTING HEMATO-ONCOLOGIE VOOR VOLWASSENEN NEDERLAND) — http://www.hovon.nl